CLINICAL TRIAL: NCT02645253
Title: A Phase I, Randomized, Single-blind, Placebo-controlled, Sequential-group, Single-center Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Ascending Doses of AZD7594 Given Once Daily as Inhaled Formulation in Healthy Japanese Men
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD7594 Inhaled Formulation in Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D3741C00005
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease COPD
Keywords: Safety; Pharmacokinetics; Pharmacodynamics; Glucocorticoid receptor modulator; Healthy male subjects
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): AZD7594 inhalation powder (200 μg) or AZD7594 placebo inhalation powder via multi-dose dry powder inhaler (DPI)
  Interventions: Drug: AZD7594 inhalation powder (200 μg); Drug: AZD7594 placebo inhalation powder
- Cohort 2 (Experimental): AZD7594 inhalation powder (400 μg) or AZD7594 placebo inhalation powder via multi-dose dry powder inhaler (DPI)
  Interventions: Drug: AZD7594 inhalation powder (400 μg); Drug: AZD7594 placebo inhalation powder
- Cohort 3 (Experimental): 1600 μg AZD7594 inhalation powder (4 x 400 μg) or AZD7594 placebo inhalation powder via multi-dose dry powder inhaler (DPI)
  Interventions: Drug: AZD7594 inhalation powder (400 μg); Drug: AZD7594 placebo inhalation powder
- Cohort 4 (Experimental): 400 μg AZD7594 pressurized inhalation suspension (2 x 200 μg inhalations) or placebo pressurized inhalation suspension via pressurized metered dose inhaler (pMDI)
  Interventions: Drug: AZD7594 pressurized inhalation suspension (200 μg); Drug: AZD7594 placebo pressurized inhalation suspension

INTERVENTIONS:
Drug: AZD7594 inhalation powder (200 μg) — 200 μg AZD7594 inhalation powder via multi-dose dry powder inhaler (DPI)
  Arms: Cohort 1
Drug: AZD7594 inhalation powder (400 μg) — Cohort 2: 400 μg AZD7594 inhalation powder via multi-dose DPI Cohort 3: 1600 μg (4 x 400 μg inhalations) AZD7594 inhalation powder via multi-dose DPI
  Arms: Cohort 2; Cohort 3
Drug: AZD7594 pressurized inhalation suspension (200 μg) — 400 μg (2 x 200 μg inhalations) AZD7594 pressurized inhalation suspension via pressurized metered dose inhaler (pMDI)
  Arms: Cohort 4
Drug: AZD7594 placebo inhalation powder — AZD7594 placebo inhalation powder via multi-dose DPI
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: AZD7594 placebo pressurized inhalation suspension — AZD7594 placebo pressurized inhalation suspension via pressurized metered dose inhaler (pMDI)
  Arms: Cohort 4

SUMMARY:
This is a randomized, single-blind, placebo-controlled, sequential-group study to assess the safety and tolerability as well as how the drug (AZD7594) affects the body (pharmacodynamics [PD]) and how the body affects the drug (pharmacokinetics [PK]) when AZD7594 is given as single and multiple ascending doses once daily by inhalation to healthy male Japanese subjects, compared with placebo (non-active drug)

DETAILED DESCRIPTION:
This is a phase I, randomized, single-blind, placebo controlled, sequential-group design study to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of AZD7594 after single and multiple ascending doses given once daily by inhalation in healthy male Japanese subjects, compared with placebo

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male Japanese subjects aged 20 to 45 years with suitable veins for cannulation or repeated venipuncture.

   A Japanese male subject is defined as being born in Japan, having both parents and four grandparents who are Japanese. The subject must not have lived outside of Japan for more than 5 years.
3. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 45 kg and no more than 100 kg inclusive.
4. Provision of signed, written and dated informed consent for optional genetic research Note: If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of investigational drug administration.
4. Any contraindication against the use of vagolytic or sympaticomimetic drugs, as judged by the investigator.
5. Any clinically significant abnormalities in clinical chemistry, hematology, urinalysis, physical examination, vital signs, electrocardiogram (ECG) or lung function results at baseline, as judged by the investigator.
6. Known Gilbert's syndrome, family history of Gilbert's syndrome or suspicion of Gilbert's syndrome based on liver function tests.
7. Use of systemic glucocorticosteroids within 6 weeks of enrollment.
8. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).
9. Known or suspected hypersensitivity to investigational product or excipients.
10. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
11. Abnormal vital signs, after 10 minutes supine rest, defined as any of the following:

    * Systolic blood pressure (BP) < 90mmHg or > 140 mmHg
    * Diastolic BP < 60mmHg or > 90 mmHg
    * Pulse rate < 40 or > 85 beats per minute (bpm)
12. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
13. Prolonged QT interval corrected for heart rate (HR) using Fridericia's formula (QTcF) > 450 ms or family history of long QT syndrome.
14. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).
15. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree AV block, or AV dissociation.
16. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation.
17. Known or suspected history of drug abuse, as judged by the investigator.
18. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
19. History of alcohol abuse or excessive intake of alcohol, as judged by the investigator.
20. Positive screen for drugs of abuse or cotinine (nicotine) at screening or admission to the unit.
21. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to ADZ7594.
22. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the investigator.
23. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of investigational drug.
24. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of investigational drug or longer if the medication has a long half-life.
25. Has received another new chemical entity (defined as a compound which has not been approved for marketing in the US) within 30 days or at least 5 half-lives (whichever is longer) of the first administration of investigational drug in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.

    Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
26. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
27. Subjects who have previously received AZD7594.
28. Involvement of any Astra Zeneca or study site employee or their close relatives.
29. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
30. Subjects who are vegans or have medical dietary restrictions.
31. Subjects who cannot communicate reliably with the investigator. It is acceptable to make use of an interpreter. The informed consent document (ICD) must be available in the Japanese language.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
32. Previous bone marrow transplant.
33. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-04-17 (Actual); Study Completion 2016-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yoon, M.D, Principal Investigator — California Clinical Trials Medical Group
Locations (1):
- Research Site, Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at PAREXEL Early Phase Clinical Unit - Los Angeles
Pre-assignment Details: Twenty-seven participants were randomized in 3 sequential cohorts. Each cohort consisted of nine participants in it. Within each cohort, 7 participants were randomly assigned to receive AZD7594 (different doses) and 2 subjects were randomly assigned to receive placebo.
Groups:
- AZD7594 200 μg: Participants received 200 μg inhaled AZD7594 via multi-dose dry powder inhaler (DPI) (1 x 200 μg inhalation)
- AZD7594 400 μg: Participants received 400 μg inhaled AZD7594 via multi-dose DPI (1 x 400 μg inhalation)
- AZD7594 1600 μg: Participants received 1600 μg inhaled AZD7594 via multi-dose DPI (4 x 400 μg inhalations).
- Palcebo: Participants received placebo
Period: Overall Study
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Palcebo
Started | 7 | 7 | 7 | 6
Completed | 7 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty-seven subjects in total were randomized to this study, 6 subjects received placebo and 21 subjects received AZD7594. All randomized subjects received treatment and completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Palcebo | Total
Number analyzed (Participants) | 7 | 7 | 7 | 6 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (5.41) | 34.1 (6.41) | 33.6 (6.43) | 35.7 (5.54) | 34.0 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 7 | 7 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD7594 by Assessment of the Number of Participants With Adverse Events
Description: To assess the safety and tolerability of single and multiple doses of AZD7594
Time Frame: At screening (Day -28, Day -02 and Day -1), Treatment period (Days 1 to 20) and Follow-up (Day 29).
Population: All subjects who received at least one dose of IMP and for whom any post-dose data were available were included in the safety analysis set.
Measure: Number; unit: Pariticpants
Groups:
- Total AZD7594: Overall number of participants who received treatment with AZD7594.
- Placebo: Participants who received placebo.
- All Subjects: Total number of participants in the study.
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Total AZD7594 | Placebo | All Subjects
Number analyzed (Participants) | 7 | 7 | 7 | 21 | 6 | 27
Pariticpants
  Any AE | 3 | 1 | 1 | 5 | 1 | 6
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE including events with outcome =death | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of IP | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Observed Maximum Plasma Concentration (Cmax)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Cmax was defined as observed maximum plasma concentration, taken directly from the individual concentration-time curve.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: The pharmacokinetic (PK) analysis set consisted of all subjects in the safety analysis set who received AZD7594 and had at least 1 measured AZD7594 plasma concentration at a scheduled PK time point post-dose, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol/L | 56.05 (22.0) | 76.93 (34.4) | 430.8 (22.4)
Statistical Analysis 1: Comparison: AZD7594 200 μg vs AZD7594 400 μg vs AZD7594 1600 μg; Test type: Superiority or Other; Linear Model; Slope = 1.02, 90% CI 2-sided [0.882 to 1.15], Standard Error of Mean 0.0785

3. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Time to Reach Maximum Plasma Concentration (Tmax)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  tmax was defined as time to reach maximum plasma concentration, taken directly from the individual concentration-time curve.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: The PK analysis set consisted of all subjects in the safety analysis set who received AZD7594 and had at least 1 measured AZD7594 plasma concentration at a scheduled PK time point post-dose, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Hours | 0.25 [0.25 to 0.98] | 0.52 [0.25 to 3.00] | 0.50 [0.25 to 4.00]

4. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Time of Last Quantifiable Analyte Concentration (AUC [0-last])
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC (0-last) was defined as the area under the plasma concentration-time curve from time zero to the time of last quantifiable analyte concentration.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
h*pmol/L | 1314 (28.2) | 2736 (12.2) | 13960 (18.2)
Statistical Analysis 1: Comparison: AZD7594 200 μg vs AZD7594 400 μg vs AZD7594 1600 μg; Test type: Superiority or Other; Linear Model; Slope = 1.14, 90% CI 2-sided [1.06 to 1.23], Standard Error of Mean 0.0503

5. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the AUC From Time Zero to 24 Hours After Dosing (AUC [0-24]).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC (0-24) was defined as area under the plasma concentration-time curve from time zero to 24 hours after dosing.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
h*pmol/L | 681.1 (11.5) | 1084 (19.4) | 6060 (18.4)

6. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the AUC From Time Zero Extrapolated to Infinity (AUC).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC was defined as area under the plasma concentration-time curve from time zero extrapolated to infinity. AUC is estimated by AUC(0-last) + Clast/λz where Clast is the last observed quantifiable concentration.
  NOTE: No results were available for participants belonging to AZD7594 2ug and AZD7594 400ug groups.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
h*pmol/L | NA (NA) — NA: Not applicable due to greater than 30% extrapolated area AUC values for most subjects were determined with >30% extrapolated area, thus were excluded from statistical analysis. | NA (NA) — NA: Not applicable due to greater than 30% extrapolated area AUC values for most subjects were determined with >30% extrapolated area, thus were excluded from statistical analysis. | 18260 (22.9)
Statistical Analysis 1: Comparison: AZD7594 200 μg vs AZD7594 400 μg vs AZD7594 1600 μg; Test type: Superiority or Other; Linear Model; Slope = 1.05, 90% CI 2-sided [0.801 to 1.31], Standard Error of Mean 0.119

7. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Terminal Elimination Rate Constant, Estimated by Log-linear Least Squares Regression of the Terminal Part of the Concentration-time Curve(Lamda z or λz).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  λz was defined as terminal elimination rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: l/h
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
l/h | 0.015573 (24.5) | 0.011058 (18.3) | 0.013862 (21.4)

8. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Half-life Associated With the Terminal Slope of a Semi-logarithmic Concentration-time Curve (t1/2λz).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  t1/2λz was defined as half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve.
  NOTE: No results were available for participants belonging to AZD7594 400ug group.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Hours | 39.88 (5.441) | NA (NA) — NA - Not applicable. When t½λz was greater than half of total sampling interval (48 hours) or percentage of AUC obtained by extrapolating area under plasma concentration-time curve (%AUCextr) was > 30%, t½λz was excluded from descriptive statistics | 43.57 (3.815)

9. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Mean Residence Time From Time Zero Extrapolated to Infinity (MRT).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  MRT was defined as Mean residence time from time zero extrapolated to infinity.
  NOTE: No results were available for participants belonging to AZD7594 200ug and AZD7594 400ug groups.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Hours | NA (NA) — NA - Not applicable. When t½λz was greater than half of the total sampling interval (48 hours) or %AUCextr was > 30%, the terminal elimination phase dependent parameter (MRT) was excluded from descriptive statistics. | NA (NA) — NA - Not applicable. When t½λz was greater than half of the total sampling interval (48 hours) or %AUCextr was > 30%, the terminal elimination phase dependent parameter (MRT) was excluded from descriptive statistics. | 65.03 (4.7)

10. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Apparent Total Body Clearance After Extravascular Administration Estimated as Dose Divided by AUC (AZD7594) (CL/F).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  CL/F was defined as apparent total body clearance after extravascular administration estimated as dose divided by AUC (AZD7594).
  NOTE: No results were available for participants belonging to AZD7594 200ug and AZD7594 400ug groups.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
L/h | NA (NA) — NA - Not applicable. When t½λz was greater than half of the total sampling interval (48 hours) or %AUCextr was > 30%, the terminal elimination phase dependent parameter (CL/F) was excluded from descriptive statistics | NA (NA) — NA - Not applicable. When t½λz was greater than half of the total sampling interval (48 hours) or %AUCextr was > 30%, the terminal elimination phase dependent parameter (CL/F) was excluded from descriptive statistics | 144.5 (22.9)

11. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration, Estimated by Dividing CL/F by Lamda z (Vz/F)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Vz/F was defined as apparent volume of distribution during the terminal phase after extravascular administration, estimated by dividing the apparent clearance (CL/F) by λz.
  NOTE: No results were available for participants belonging to AZD7594 200ug and AZD7594 400ug groups.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Litres | NA (NA) — NA - Not applicable. When t½λz was greater than half of the total sampling interval (48 hours) or %AUCextr was > 30%, the terminal elimination phase dependent parameter (Vz/F) was excluded from descriptive statistics | NA (NA) — NA - Not applicable. When t½λz was greater than half of the total sampling interval (48 hours) or %AUCextr was > 30%, the terminal elimination phase dependent parameter (Vz/F) was excluded from descriptive statistics | 9297 (24.1)

12. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Cmax Divided by the Dose Administered (Cmax/D).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Cmax/D was defined as observed maximum plasma concentration divided by the dose administered.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pmol/L)/umol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
(pmol/L)/umol | 169.9 (22.0) | 116.7 (34.4) | 163.2 (22.4)

13. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the AUC Divided by the Dose Administered (AUC/D).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC/D was defined as Area under the plasma concentration-time curve from time zero extrapolated to infinity divided by the dose administered.
  NOTE: No results were available for participants belonging to AZD7594 200ug and AZD7594 400ug groups.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pmol*h/L)/umol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
(pmol*h/L)/umol | NA (NA) — NA - Not available For 6 participants, %AUCextr was > 30%. Hence, values were excluded from descriptive statistics. | NA (NA) — NA - Not available NA - Not available For all participants, %AUCextr was > 30%. Hence, values were excluded from descriptive statistics. | 6918 (22.9)

14. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the AUC(0-24) Divided by the Dose Administered (AUC(0-24)/D)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC(0-24)/D was defined as area under the plasma concentration-time curve from time zero to 24 hours after dosing divided by the dose administered.
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pmol*h/L)/umol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
(pmol*h/L)/umol | 2064 (11.5) | 1645 (19.4) | 2295 (18.4)

15. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Observed Minimum Plasma Concentration (Cmin)
Description: Cmin was defined as observed minimum plasma concentration, taken directly from the individual concentration-time curve
Time Frame: Days 5 to 15: Pre-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol/L
  Day 5 - Pre-dose | NA (NA) — NA: Not applicable 6 participants were in below lower limit of quantification (10 pmol/L) category | 16.27 (13.13) | 68.91 (21.55)
  Day 5 - 1 hour | 59.81 (27.60) | 77.10 (26.92) | 404.2 (22.74)
  Day 6 - Pre-dose | 29.35 (17.83) | 47.75 (20.76) | 252.2 (24.53)
  Day 7 - Pre-dose | 41.59 (10.33) | 76.91 (16.27) | 369.0 (20.88)
  Day 8 - Pre-dose | 51.99 (12.29) | 92.18 (18.17) | 458.4 (22.39)
  Day 8 - 1 hour | 106.4 (19.69) | 162.3 (20.93) | 793.0 (26.60)
  Day 9 - Pre-dose | 60.37 (16.48) | 108.2 (25.11) | 548.3 (25.72)
  Day 10 - Pre-dose | 61.88 (21.52) | 119.3 (31.01) | 554.2 (23.65)
  Day 11 - Pre-dose | 68.39 (19.83) | 136.3 (26.20) | 623.5 (21.10)
  Day 12 - Pre-dose | 78.39 (9.019) | 142.6 (30.88) | 603.8 (16.84)
  Day 12 - 1 hour | 139.5 (8.216) | 219.8 (26.21) | 925.8 (16.61)
  Day 13 - Pre-dose | 79.31 (12.92) | 145.5 (38.15) | 698.3 (19.89)
  Day 14 - Pre-dose | 77.04 (7.165) | 147.0 (34.87) | 718.4 (23.65)
  Day 15 - Pre-dose | 82.40 (13.30) | 151.9 (35.42) | 694.9 (11.67)

16. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Cmax at Steady State (Css,Max).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Css,max was defined as observed maximum plasma concentration at steady state, taken directly from the individual concentration-time curve.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol/L | 164.3 (14.0) | 261.2 (37.0) | 1206 (14.7)
Statistical Analysis 1: Comparison: AZD7594 200 μg vs AZD7594 400 μg vs AZD7594 1600 μg; Test type: Superiority or Other; Linear Model; Slope = 0.979, 90% CI 2-sided [0.870 to 1.09], Standard Error of Mean 0.0633

17. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Cmin at Steady State (Cmin, ss)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Cmin, ss was defined as observed minimum concentration, taken directly from the individual concentration-time curve.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol/L | 82.15 (12.8) | 140.6 (38.5) | 600.0 (27.0)

18. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Average Concentration Over One Dosing Interval (Cav)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Cav was defined as average concentration over one dosing interval.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol/L | 101.1 (13.4) | 183.7 (33.4) | 867.8 (13.2)

19. Secondary Outcome: Rate and Extent of Absorption of AZD7594 (Inhalation/ Administration Via DPI) by Assessment of the Tmax at Steady State (Tss,Max).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  tss,max was defined as Time to reach maximum concentration, taken directly from the individual concentration-time curve.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Hours | 0.25 [0.25 to 4.02] | 1.50 [0.25 to 8.00] | 1.50 [0.25 to 4.00]

20. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the AUC(0-last)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC(0-last) was defined as Area under the plasma concentration-time curve from time zero to the time of the last quantifiable analyte concentration.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol*h/L | 6136 (16.2) | 11490 (36.9) | 54120 (11.5)

21. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of AUC(0-24)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC(0-24) was defined as area under the plasma concentration-time curve from time zero to 24 hours after dosing
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol*h/L | 2426 (13.4) | 4409 (33.4) | 20830 (13.2)
Statistical Analysis 1: Comparison: AZD7594 200 μg vs AZD7594 400 μg vs AZD7594 1600 μg; Test type: Superiority or Other; Linear Model; Slope = 1.05, 90% CI 2-sided [0.951 to 1.14], Standard Error of Mean 0.0552

22. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Css,Max Divided by the Dose Administered (Css,Max/D).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Css,max/D was defined as observed maximum plasma concentration divided by the dose administered.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pmol/L)/umol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
(pmol/L)/umol | 498.0 (14.0) | 396.4 (37.0) | 456.9 (14.7)

23. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment AUC(0-24)/D.
Description: Assessment of the plasma PK following a single dose of AZD7594.
  AUC(0-24)/D was defined as the area under the plasma concentration-time curve from time zero to 24 hours after dosing divided by the dose administered.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (pmol*h/L)/umol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
(pmol*h/L)/umol | 7351 (13.4) | 6691 (33.4) | 7889 (13.2)

24. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of Lamda z (λz)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  λz was defined as terminal elimination rate constant, estimated by log-linear least.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: l/hour
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
l/hour | 0.013393 (19.8) | 0.011465 (38.8) | 0.010660 (27.4)

25. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of t1/2λz.
Description: Assessment of the plasma PK following a single dose of AZD7594.
  t1/2λz was defined as half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve.
  Participant count analyzed = 1
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Hours | NA (NA) — NA - Not applicable When Rsq_adj (regression co-efficient adjusted for λz) was < 0.7 or estimated t1/2λz was greater than half of the total sampling interval (48 hours), t½λz was excluded from descriptive statistics | NA (NA) — NA - Not applicable When Rsq_adj (regression co-efficient adjusted for λz) was < 0.7 or estimated t1/2λz was greater than half of the total sampling interval (48 hours), t½λz was excluded from descriptive statistics | NA (NA) — NA - Not applicable When Rsq_adj (regression co-efficient adjusted for λz) was < 0.7 or estimated t1/2λz was greater than half of the total sampling interval (48 hours), t½λz was excluded from descriptive statistics

26. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Peak Trough Fluctuation (%Fluctuation).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Peak trough fluctuation calculated as [100*(Css,max- Css,min)/Cav].
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: The pharmacodynamics analysis set will include all subjects who receive at least 1 dose of IMP and for whom it is possible to calculate the cortisol AUEC on Day -1, Day 1 and/or Day 16 and with no major protocol deviations considered to impact on the analysis of the PD (cortisol, plasma DHEAS and osteocalcin) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of fluctuation
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Percentage of fluctuation | 80.12 (23.8) | 64.61 (21.8) | 68.08 (21.0)

27. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Accumulation Ratio Calculated as AUC(0-24) on Day 16/AUC (0-24) on Day 1 (RAC).
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Accumulation ratio calculated as AUC(0-24) on Day 16/AUC(0-24) on Day 1.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Ratio | 3.562 (15.7) | 4.067 (43.7) | 3.437 (7.3)

28. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Temporal Change Parameter (TCP)
Description: Assessment of the plasma PK following a single dose of AZD7594.
  Temporal change parameter, calculated as AUC(0-24) [Day 16]/AUC [Day 1].
  NOTE: No results were available for participants belonging to AZD7594 200ug and AZD7594 400ug groups.
Time Frame: Day 16: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Ratio | NA (NA) — NA - Not available For all participants, AUC value on Day 1 could not be reliably determined. Hence, values were excluded from descriptive statistics | NA (NA) — NA - Not available For all participants, AUC value on Day 1 could not be reliably determined. Hence, values were excluded from descriptive statistics | 1.147 (7.7)

29. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Amount of AZD7594 Excreted Into the Urine From Time t1 to t2 (Ae [t1-t2])
Description: Assessment of the urine PK following a single dose of AZD7594.
  Ae (t1-t2) was defined as the amount of AZD7594 excreted into the urine from time t1 to t2.
Time Frame: Day 1 predose spot-collection and interval collection up to 96 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol
  0-6h | 1.856 (4.910) | 6.738 (9.751) | 55.64 (58.01)
  6-12h | 1.434 (3.795) | 5.031 (6.645) | 73.15 (53.23)
  12-24h | 1.893 (5.008) | 1.907 (5.046) | 73.13 (50.96)
  24-48h | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | 107.9 (76.97)
  48-72h | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | 72.43 (58.77)
  72-96h | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | 48.95 (48.49)

30. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Cumulative Amount of AZD7594 Excreted From Time Zero to the Last Sampling Interval (Ae [0-last])
Description: Assessment of the urine PK following a single dose of AZD7594.
  Ae(0-last) was defined as Cumulative amount of AZD7594 excreted from time zero to the last sampling interval.
Time Frame: Day 1 predose spot-collection and interval collection up to 96 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pmol
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
pmol
  0-6h | 1.856 (4.910) | 6.738 (9.751) | 55.64 (58.01)
  0-12h | 3.290 (8.705) | 11.77 (15.25) | 128.8 (83.03)
  0-24h | 5.183 (13.71) | 13.68 (17.07) | 201.9 (117.9)
  0-48h | 5.183 (13.71) | 13.68 (17.07) | 309.9 (175.6)
  0-72h | 5.183 (13.71) | 13.68 (17.07) | 382.3 (219.7)
  0-96h | 5.183 (13.71) | 13.68 (17.07) | 431.2 (262.2)

31. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Percentage of Dose Excreted Unchanged Into the Urine From Time Zero to the Last Measured Time Point for an AZD7594, Estimated by Dividing Ae(0-last) by Dose (fe(0-last)%)
Description: Assessment of the urine PK following a single dose of AZD7594.
  fe(0-last)% was defined as Percentage of dose excreted unchanged into the urine from time zero to the last measured time point for an AZD7594, estimated by dividing Ae(0-last) by dose.
Time Frame: Day 1 predose spot-collection and interval collection up to 96 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of dose excreted unchanged
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
Percentage of dose excreted unchanged
  0-6h | 0.0005623 (0.001488) | 0.001022 (0.001480) | 0.002108 (0.002197)
  6-12h | 0.0004346 (0.001150) | 0.0007634 (0.001008) | 0.002771 (0.002016)
  12-24h | 0.0005736 (0.001518) | 0.0002894 (0.0007657) | 0.002770 (0.001930)
  24-48h | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | 0.004088 (0.002915)
  48-72h | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | 0.002743 (0.002226)
  72-96h | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | NA (NA) — NA - Not available Participants concentration values were below lower limit of quantitation (10 pmol/L) category | 0.001854 (0.001837)

32. Secondary Outcome: Rate and Extent of Absorption of AZD7594 by Assessment of the Renal Clearance, Estimated by Dividing Ae(0-96) by AUC(0-96) (CLR)
Description: Assessment of the urine PK following a single dose of AZD7594.
  CLR was defined as the renal clearance, estimated by dividing Ae(0-96) by AUC(0-96).
Time Frame: Day 1 predose spot-collection and interval collection up to 96 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg
Number analyzed (Participants) | 7 | 7 | 7
L/h | NA (NA) — NA - Not available Since, %AUCextr was > 30%, values were excluded from descriptive statistics | NA (NA) — NA - Not available Since, %AUCextr was > 30%, values were excluded from descriptive statistics | 0.02329 (98.8)

33. Secondary Outcome: Pharmacodynamic Analysis of AZD7594 by Assessment of the Area Under the Effect Curve for Plasma Cortisol From Time Zero to 24 Hours After Dosing (AUEC [0-24]).
Description: Assessment of the plasma pharmacodynamics (PD) effects of AZD7594 after single and multiple ascending inhaled doses.
  AUEC(0-24) was defined as area under the effect curve for plasma cortisol from time zero to 24 hours after dosing.
Time Frame: Day -1 (- 24 hours predose) up to 24 hours postdose; Day 1 and Day 16
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: min*nmol/L
Groups:
- Placebo: Participants received placebo.
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 6
min*nmol/L
  Day -1 | 294273.817 (66921.717) | 286677.610 (41429.744) | 298827.031 (57082.835) | 275402.666 (42811.506)
  Day 1 | 268228.553 (34086.352) | 274458.997 (36894.669) | 264104.101 (47619.269) | 256226.560 (48755.915)
  Day 16 | 253767.846 (11407.064) | 249097.459 (46925.914) | 213505.523 (40857.201) | 273268.869 (57797.995)
Statistical Analysis 1: Comparison: AZD7594 200 μg vs Placebo; Test type: Superiority or Other; ANCOVA; Ratio of Geometric LS mean (%) = 102.99, 95% CI 2-sided [86.88 to 122.09] — Day 1/ Day -1
Statistical Analysis 2: Comparison: AZD7594 200 μg vs Placebo; Test type: Superiority or Other; ANCOVA; Ratio of Geometric LS mean (%) = 91.82, 95% CI 2-sided [77.32 to 109.04] — Day 16 / Day -1
Statistical Analysis 3: Comparison: AZD7594 400 μg vs Placebo; Test type: Superiority or Other; ANCOVA; Ratio of Geometric LS mean (%) = 105.92, 95% CI 2-sided [89.40 to 125.49] — Day 1 / Day -1
Statistical Analysis 4: Comparison: AZD7594 400 μg vs Placebo; Test type: Superiority or Other; ANCOVA; Ratio of Geometric LS mean (%) = 89.44, 95% CI 2-sided [75.35 to 106.16] — Day 16 / Day -1
Statistical Analysis 5: Comparison: AZD7594 1600 μg vs Placebo; Test type: Superiority or Other; ANCOVA; Ratio of Geometric LS mean (%) = 99.82, 95% CI 2-sided [84.12 to 118.46] — Day 1 / Day -1
Statistical Analysis 6: Comparison: AZD7594 1600 μg vs Placebo; Test type: Superiority or Other; ANCOVA; Ratio of Geometric LS mean (%) = 75.38, 95% CI [63.40 to 89.61] — Day 16 / Day -1

34. Secondary Outcome: Pharmacodynamic Analysis of AZD7594 by Assessment of Plasma Concentration of Dehydroepiandrosterone Sulphate (DHEAS)
Description: Assessment of the plasma PD following a single dose of AZD7594
Time Frame: Day 1 (predose) and Day 16 (24 hours postdose)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 6
μmol/L
  Result: Day 1 / pre-dose | 6.716 (1.405) | 7.380 (2.429) | 6.747 (2.936) | 6.280 (1.829)
  Result: Day 17 / 24 h | 6.104 (0.862) | 6.250 (1.005) | 7.125 (2.708) | 6.392 (2.179)

35. Secondary Outcome: Pharmacodynamic Analysis of AZD7594 by Assessment of Plasma Concentration of Osteocalcin
Description: Assessment of the plasma PD following a single dose of AZD7594
Time Frame: Day 1 (predose) and Day 16 (24 hours postdose)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Placebo
Number analyzed (Participants) | 7 | 7 | 7 | 6
μg/L
  Day 1 / pre-dose | 21.31 (17.22) | 23.13 (10.02) | 20.01 (5.77) | 22.92 (20.13)
  Day 17 / 24 h | 17.81 (8.55) | 19.66 (11.56) | 13.37 (8.26) | 17.03 (5.60)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were recorded from the signing of informed consent and adverse events (AEs) were recorded from randomization until the final follow-up visit.
Description: An AE is an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. AEs which met the "Definitions of Serious Adverse Event" defined in the clinical study protocol were regarded as SAEs.
Groups:
- Total AZD7594: Overall number of subjects who received AZD7594 therapy.
- All Subjects: Overall number of subjects who participated in the study.
Arm/Group | AZD7594 200 μg | AZD7594 400 μg | AZD7594 1600 μg | Palcebo | Total AZD7594 | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/6 | 0/21 | 0/27
Other Adverse Events (participants affected / at risk) | 3/7 | 1/7 | 1/7 | 1/6 | 5/21 | 6/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7594 200 μg (N=7) | AZD7594 400 μg (N=7) | AZD7594 1600 μg (N=7) | Palcebo (N=6) | Total AZD7594 (N=21) | All Subjects (N=27)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.